CLINICAL TRIAL: NCT04564885
Title: A Multicenter, Prospective, Randomized, Clinical Trial Comparing the Safety and Effectiveness of the BAGUERA C Cervical Disc Prosthesis to the Mobi-C® Cervical Disc for the Treatment of Patients With Symptomatic Cervical Disc Disease at Two Contiguous Levels
Brief Title: A Clinical Trial Comparing the BAGUERA C to the Marketed Mobi-C® for the Treatment of Cervical Disc Disease at 2 Contiguous Levels
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Spineart USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT-20-002-001
Record Dates: First submitted 2020-09-21; First posted 2020-09-25 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cervical Disc Disease
Keywords: radiculopathy; myeloradiculopathy
MeSH Terms: conditions — Radiculopathy

STUDY DESIGN:
Who Masked: Participant
Masking Description: participants will not be told their treatment group prior to surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- BAGUERA®C (Experimental): surgical placement of the BAGUERA®C Cervical Disc Prosthesis at 2 contiguous levels
  Interventions: Device: BAGUERA®C Cervical Disc Prosthesis
- Mobi-C® (Active Comparator): surgical placement of the Mobi-C® Cervical Disc at 2 contiguous levels
  Interventions: Device: Mobi-C Cervical Disc

INTERVENTIONS:
Device: BAGUERA®C Cervical Disc Prosthesis — surgery
  Arms: BAGUERA®C
Device: Mobi-C Cervical Disc — surgery
  Arms: Mobi-C®

SUMMARY:
The proposed investigation is a multi-center, prospective, randomized, controlled comparison of the BAGUERA®C to the control, a similar, legally marketed total disc replacement device in subjects with symptomatic cervical disc disease (SCDD) at two contiguous levels. Subjects will be randomized in a 2:1 ratio to the two-level BAGUERA®C Cervical Disc Prosthesis (investigational group) or to the two-level Mobi-C® Cervical Disc (control group). Subjects enrolled in the study will be evaluated pre-operatively, at the time of surgery, discharge, and at 6 weeks, 3, 6, 12, and 24 months and then annually until 7 years post-surgery.

ELIGIBILITY:
Inclusion Criteria

In order to be eligible to participate in this study, subjects must meet all of the following criteria:

1. Male or female; skeletally mature; age 22-69 years, inclusive.
2. Diagnosis of radiculopathy or myeloradiculopathy of the cervical spine, with pain, paresthesia or paralysis in a specific nerve root distribution C3 through C7, including at least one of the following:

   1. Neck and/or arm pain (at least 40 mm on the 100 mm visual analogue scale [VAS] scale).
   2. Decreased muscle strength of at least one level on the clinical evaluation 0 to 5 scale.
   3. Abnormal sensation including hyperesthesia or hypoesthesia; and/or
   4. Abnormal reflexes.
3. Symptomatic cervical disc disease (SCDD) at two contiguous levels from C3 to C7.
4. Radiographically determined pathology at the level to be treated correlating to primary symptoms including at least one of the following:

   1. Decreased disc height on radiography, computed tomography (CT), or magnetic resonance imaging (MRI) in comparison to a normal adjacent disc.
   2. Degenerative spondylosis on CT or MRI.
   3. Disc herniation on CT or MRI.
5. NDI Score of ≥ 30% (raw score of ≥15/50).
6. Preoperative neck or arm pain ≥ 40 (out of 100) on Preoperative Neck and Arm Pain Questionnaire.
7. Unresponsive to non-operative, conservative treatment (including but not necessarily limited to: rest, heat, electrotherapy, physical therapy, chiropractic care and/or analgesics) for:

   1. Approximately six weeks from radiculopathy or myeloradiculopathy symptom onset; or
   2. Have the presence of progressive symptoms or signs of nerve root/spinal cord compression despite continued non-operative conservative treatment.
8. Appropriate for treatment using an anterior surgical approach, including having no prior surgery at the operative level and no prior cervical fusion or cervical artificial disc procedure at any level.
9. Medically cleared for surgery.
10. Physically and mentally able and willing to comply with the Protocol, including the ability to read and complete required forms and willing and able to adhere to the scheduled follow-up visits and requirements of the Protocol.
11. Written informed consent provided by Subject

Exclusion Criteria

Patients are not permitted to enroll in the two-level BAGUERA®C study if they meet any of the following exclusion criteria:

1. Have an active systemic infection or infection at the operative site.
2. Have a history of or anticipated treatment for active systemic infection, including HIV or Hepatitis C.
3. More than one immobile vertebral level between C1 to C7 from any cause including but not limited to congenital abnormalities and osteoarthritic "spontaneous" fusions.
4. Previous trauma to the C3 to C7 levels resulting in significant bony or disco-ligamentous cervical spine injury.
5. Had any prior spine surgery at the operative level(s).
6. Had a prior fusion or artificial disc procedure at any cervical level.
7. Axial neck pain alone in the absence of other symptoms of radiculopathy or myeloradiculopathy.
8. Disc height less than 3 mm as measured from the center of the disc in a neutral lateral position.
9. Radiographic confirmation of severe facet joint degeneration or confirmed clinical evidence that facet joint degeneration is a major contributor to the subject's pain.
10. Have osteoporosis or osteopenia, defined as a DEXA bone density measured T-score of ≤ -1.5 (i.e. -1.6, -1.7, etc.). A DEXA performed within 24 months of the surgery date may be used to determine eligibility. For subjects without a DEXA within 24 months of the surgery date a score of ≥ 6 on either the SCORE or MORES requires a DEXA to determine eligibility. Note: The SCORE (Simple Calculated Osteoporosis Risk Estimation) form should be administered if the subject is female. The MORES (Male Osteoporosis Risk Estimation Score) form should be administered if the subject is male.
11. Have Paget's disease, osteomalacia or any other metabolic bone disease other than osteoporosis, which is addressed above.
12. Severe diabetes mellitus requiring daily insulin management.
13. Have an active malignancy that includes a history of any invasive malignancy (except non-melanoma skin cancer), unless the subject was treated with curative intent and there had been no clinical signs or symptoms of the malignancy for at least five years.
14. Symptomatic SCDD or significant cervical spondylosis at more than two levels.
15. Spondylolysis.
16. Marked cervical instability on resting lateral or flexion-extension radiographs demonstrated by:

    1. Translation ≥ 3.5 mm, and/or
    2. Greater than 11° angular difference to that of either adjacent level.
17. Known allergy to Titanium, Vanadium, Aluminum, Cobalt, Chromium, Molybdenum or Polyethylene.
18. Segmental angulation of greater than 11° at treatment or adjacent levels.
19. Pregnant at time of enrollment, or with plans to become pregnant within the next three years.
20. Have rheumatoid arthritis, lupus, or other autoimmune disease that affect the musculoskeletal system.
21. Congenital bony and/or spinal cord abnormalities that affect spinal stability.
22. Have diseases or conditions that would preclude accurate clinical evaluation (e.g. neuromuscular disorders, confirmed fibromyalgia, etc.).
23. Concomitant conditions requiring daily, high-dose oral and/or inhaled steroids. High dose steroid use is defined as:

    1. Daily, chronic use of oral steroids of 5 mg/day or greater.
    2. Daily, chronic use of inhaled corticosteroids (at least twice per day).
    3. Use of short-term (less than 10 days) oral steroids at a daily dose greater than 40mg within one month of the study procedure.
24. Have current or recent history of substance abuse (alcoholism and/or narcotic addiction) requiring intervention.
25. Severe Obesity, as defined by National Institutes of Health (NIH) Clinical Guidelines Body Mass Index (BMI) > 40).
26. Use of any investigational drug or other investigational medical device within the last 30 days prior to surgery.
27. Taking medications known to interfere with bone/soft tissue healing (e.g., high-dose oral and/or inhaled steroids, immunosuppressant medication, chemotherapeutic agents). High dose steroid use is defined as part of Exclusion Criterion #23.
28. Currently pursuing litigation (defined as litigation that will likely influence the patient's ability or willingness to accurately report their treatment outcomes) related to the neck or cervical spine injury.
29. Current history of heavy nicotine use (e.g. more than one pack of cigarettes per day).
30. Circumstances that may interfere with completion of follow-up examinations, including location of residence.
31. Belong to a vulnerable population (e.g., prisoner, wards of the court or developmentally disabled).
32. Currently experiencing an acute or chronic episode of confirmed specific mental illness (psychosis, major affective disorder, or schizophrenia), or manifesting physical symptoms without a diagnosable medical condition to account for the symptoms, which may indicate symptoms of psychological rather than physical origin.
33. Have an uncontrolled seizure disorder.
34. Received cervical spine epidural steroids within 14 days prior to surgery.

Ages: 22 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-03-02 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2030-04 (Estimated)

PRIMARY OUTCOMES:
Neck Disability Index | 24 month follow-up visit
  at least a 15 percentage point improvement (decrease) from baseline on a 0 - 100% scale
Maintenance or improvement in neurological status | 24 month follow-up visit
  pre and post-op neurological examination to determine maintenance or improvement
No secondary surgical intervention per protocol definition | 24 month follow-up visit
  any revision, removal, re-operation, or supplemental fixation at the index level
Procedure or device related serious adverse events | 24 month follow-up visit
  No serious adverse event(s) confirmed as device or procedure related as adjudicated by the Clinical Events Committee

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - MORE Foundation, Phoenix, Arizona
  - Desert Institute for Spine Care, Scottsdale, Arizona
  - BEEL Medical, Laguna Hills, California
  - Orange County Neurosurgical Associates, Mission Viejo, California
  - UCI Health, Orange, California
  - Eisenhower Medical Center, Rancho Mirage, California
  - The Spine Institute, Center for Spine Restoration, Santa Monica, California
  - Institute for Neuro Innovation, West Hills, California
  - Vail-Summit Orthopaedics and Neurosurgery, Vail, Colorado
  - Hartford Health CT Orthopaedics, Hamden, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Legacy Brain & Spine, Atlanta, Georgia
  - Midwest Orthopedics at Rush, Chicago, Illinois
  - NorthShore, Evanston, Illinois
  - Indiana Spine Group, Carmel, Indiana
  - Ortho NorthEast, Fort Wayne, Indiana
  - Orthopaedic Institute of Western Kentucky, Paducah, Kentucky
  - Spine Institute of Louisiana Foundation, Shreveport, Louisiana
  - Carolina Neurosurgery and Spine Associates, Charlotte, North Carolina
  - The Ohio State University - Dept of Orthadedics, Columbus, Ohio
  - Oregon Spine Care, Tualatin, Oregon
  - Neurosurgical Associates of Lancaster, Lancaster, Pennsylvania
  - Center for Sports Medicine & Orthopedics, Chattanooga, Tennessee
  - St. David's Healthcare, Austin, Texas
  - The Disc Replacement Center, Salt Lake City, Utah
  - Swedish Neuroscience, Swedish Spine Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No